CLINICAL TRIAL: NCT00309868
Title: A Study of the Acute Hemodynamic and Myocardial Effects of Nesiritide in Diastolic Heart Failure.
Brief Title: Study of Nesiritide in Diastolic Heart Failure.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Semigran, Medical Director , Heart Failure and Cardiac Transplantation, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-p-001736
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Diastolic Heart Failure
Keywords: heart catheterization; echocardiogram; nesiritide
MeSH Terms: conditions — Heart Failure, Diastolic

INTERVENTIONS:
Drug: neseritide
  Other Names: BNP

SUMMARY:
We hypothesize that nesiritide will have favorable effect in decreasing heart filling pressures and echocardiogram studies.

DETAILED DESCRIPTION:
In previous studies, patients with systolic heart failure were given nesiritide and had reduced heart filling pressures. The FDA has approved nesiritide for these patients.

Between one-third and one-half of patients with heart failure have diastolic heart failure. Few of these patients have been studied while receiving nesiritide.

A study is needed to test nesiritide on this specific type of heart failure.

Patients will undergo a heart catheterization and heart biopsy. Patients will then be transferred to the intensive care unit for monitoring. An echocardiogram will be obtained, followed by an infusion of nesiritide for 24 hours. At the completion of the infusion, a repeat echocardiogram will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Elevated heart filling pressure. Ejection fraction >45%. Blood pressure >90. Physician feels that the patient needs intravenous medication for heart failure.

-

Exclusion Criteria:

Patients receiving intravenous medication. Patients with significant heart disease or who are unstable. Patients with kidney failure or severe heart valve disease.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2002-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc J S, MD, Principal Investigator — Massachusetts General Hospital